CLINICAL TRIAL: NCT02874885
Title: Circulating Tumor Elements in Patients With Rectal Cancer
Brief Title: Circulating Tumor Cells in Patients With Locally Advanced Rectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA13-0547; NCI-2020-07460 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA13-0547 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Rectal Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Rectosigmoid Adenocarcinoma; Recurrent Rectal Adenocarcinoma; Recurrent Rectosigmoid Carcinoma; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients and healthy participants undergo collection of blood sample at baseline. Patients may also undergo collection of blood sample collections during tumor surgery, 4 weeks after surgery or after completion of treatment if you are not surgery, 8 weeks after the last dose of chemotherapy, 1 year after surgery or 1 year after completion of treatment if not having surgery, 2 years after surgery or 2 years after completion of treatment if not having surgery, and within 6 years after treatment or at the end of the 6 year follow-up if the disease gets worse with treatment or comes back.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample

SUMMARY:
This study looks at the level of circulating tumor elements (cancer cells or DNA pieces floating in the blood) and how it may be related to how the tumor responds to standard treatment in patients with rectal cancer that has spread to nearby tissue or lymph nodes (locally advanced). Researchers will also compare the level and genetic characteristics of circulating tumor elements between individuals with rectal cancer and healthy individuals to understand how they may change over time. Information from this study may help researchers better understand rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the rate of circulating tumor elements (CTE), including but not limited to circulating tumor cells and circulating tumor deoxyribonucleic acid (DNA) detection in patients with locally advanced rectal cancer (LARC), relative to other stages.

II. To assess changes in detected CTEs associated with neoadjuvant therapy in patients with LARC.

III. To correlate CTEs with neoadjuvant treatment response as an indicator of disease risk.

OUTLINE:

Patients and healthy participants undergo collection of blood sample at baseline. Patients may also undergo collection of blood sample collections during tumor surgery, 4 weeks after surgery or after completion of treatment if you are not surgery, 8 weeks after the last dose of chemotherapy, 1 year after surgery or 1 year after completion of treatment if not having surgery, 2 years after surgery or 2 years after completion of treatment if not having surgery, and within 6 years after treatment or at the end of the 6 year follow-up if the disease gets worse with treatment or comes back.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY SUBJECT: No known diagnosis of colorectal cancer (CRC) or any other type of cancer for the last 10 years.(basal cell skin cancer is allowed). Subjects will be asked about their cancer history and a verbal confirmation is required
* Any patient with diagnosis of rectal (or rectosigmoid) adenocarcinoma, including:

  * Patients with primary disease with or without neoadjuvant therapy; OR
  * Patients with recurrent disease with or without neoadjuvant therapy; OR
  * Patients with metastatic disease with or without prior treatment
* No known current diagnosis of other invasive cancer; if prior diagnosis of other cancer, he/she has been free from cancer for >= 3 years and is on no active treatment
* Adequate mental and language capacity to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants and patients diagnosed with rectal (or rectosigmoid) adenocarcinoma at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment naive locally advanced rectal cancer (LARC) patients with circulating tumor cells (CTC) | Baseline up to 6 years
  The proportion of patients with any CTC will be calculated with a 95% confidence interval (CI). Additionally, the actual CTC count will be plotted with a box-plot. Proportions of patients with 2 or more, and 3 or more CTCs will be calculated. Will also explore correlations between the presence of 1 or more CTC and primary tumor characteristics using Chi-Squared or Fischer's exact tests as appropriate.
Change in circulating tumor cells status | Baseline and 8 weeks after completion of treatment
  A McNemar's test will be used to test whether neoadjuvant therapy (NEO) provided any improvement in the proportion of patients with any CTC. The CTC counts at baseline versus 8 weeks after completion of treatment will be compared with a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Qian N You, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org